CLINICAL TRIAL: NCT04578613
Title: A Randomized, Controlled, Open, Multicenter Phase 3 Study to Evaluate ICP-022 Versus Chlorambucil Combined With Rituximab for Primary Treatment of Chronic Lymphocytic Leukemia(CLL)/ Small Lymphocytic Lymphoma(SLL)
Brief Title: ICP-022 Versus Chlorambucil Combined With Rituximab in the Treatment of Untreated CLL/SLL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00111
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Chlorambucil; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICP-022 (Experimental): ICP-022 will be orally administered until disease progression or unacceptable toxicity.
  Interventions: Drug: ICP-022
- Chlorambucil combined with Rituximab (Active Comparator): Chlorambucil orally administered and Rituximab via IV infusion for 6 cycles.
  Interventions: Drug: Chlorambucil; Drug: Rituximab

INTERVENTIONS:
Drug: ICP-022 — ICP-022 at a dose of 150mg, QD
  Arms: ICP-022
Drug: Chlorambucil — 0.5 mg/kg body weight orally on Day 1 and Day 15 of Cycles 1-6
  Arms: Chlorambucil combined with Rituximab
Drug: Rituximab — 375 mg/m2 IV infusion on Day 1 of Cycle 1. 500 mg/m2 IV infusion on Day 1 for each of subsequent cycles (Cycles 2-6)
  Arms: Chlorambucil combined with Rituximab

SUMMARY:
This is a randomized, multicenter, open-label, Phase 3 study to evaluate the efficacy and safety of ICP-022 versus Chlorambucil plus Rituximab in subjects with Previously Untreated Chronic Lymphocytic Leukemia.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, age ≥65 years old or age >18 years old or <65 years old, age >18 years old or <65 years old shall meet any of the following criteria simultaneously: A.Disease accumulation score (CIRS) > 6;B. Creatinine clearance at 30-69 mL/ min (Cockcroft-Gault assessment)
2. Enhanced computed tomography/magnetic resonance imaging (CT/MRI) detection had measurable lesions: at least one lymph node had a maximum axis of more than 1.5 cm and had a measurable vertical dimension
3. ECOG physical strength score is 0-2.
4. Expected survival time >6 months.
5. Voluntary written informed consent prior to screening.

Key Exclusion Criteria:

1. Patients with stroke or intracranial hemorrhage in the first 6 months were randomly assigned.
2. Hypersensitivity to ICP-022, nitrogen mustard benzoate, rituximab or any other component of the applicable study drug.
3. Any mental or cognitive impairment that may limit their understanding of the informed consent, their implementation and their compliance with the study.
4. Pregnant and lactating women, or subjects of childbearing age who do not want to use contraception within 180 days from the end of the study period to the end of the study period.
5. Conditions in which a potentially life-threatening illness or severe organ dysfunction is not considered appropriate by the investigator.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 5 years
  Progress-free survival (PFS) was evaluated by the independent review board (IRC) against the IWCLL2018 criteria (Hallek et al., 2018) and the revised lymphoma mitigation assessment criteria (Cheson et al., 2014).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 5 years
Duration Of Response (DOR) | Up to 5 years
Overall Survival (OS) | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (56):
- China (56):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Congqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Cancer Prevention and Treatment Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Hebei Medical University Second Hospital, Shijiazhuang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The first Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Province Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of WuHan University, Wuhan, Hubei
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Yichang First People's Hospital, Yichang, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Subei People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Binzhou Medical College, Binzhou, Shandong
  - Shandong Cancer Hospita, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi´an Jiaotong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The first Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - Shaoyifu Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No